CLINICAL TRIAL: NCT05351255
Title: Motor Learning After Cerebellar Damage: The Role of the Primary Motor Cortex
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Amanda Therrien, PhD, Principal Investigator, Albert Einstein Healthcare Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AEHN-IRB-2022-881; P2CHD086844 (NIH)
Record Dates: First submitted 2022-04-06; First posted 2022-04-28 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-01

CONDITIONS: Cerebellar Ataxia
MeSH Terms: conditions — Cerebellar Ataxia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rTMS Intervention (Experimental): In aim 2 of the study, participants receive a repetitive transcranial magnetic stimulation intervention called theta burst stimulation (TBS) to study its effect on motor learning behavior. All participants will complete 3 sessions in which they will receive continuous TBS, intermittent TBS, or sham TBS before completing a behavioral motor learning task. The order of TBS sessions will be counter-balanced across participants.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Aim 2 of the study includes an intervention where participants receive a repetitive TMS protocol called theta burst stimulation (TBS) to study its effect on motor learning behavior.

SUMMARY:
This study will determine (1) whether baseline inhibitory activity in the primary motor cortex can predict motor learning ability in individuals with cerebellar degeneration, and (2) whether modulating primary motor cortex activity with non-invasive brain stimulation alters motor learning ability in this population.

DETAILED DESCRIPTION:
Cerebellar damage causes the disabling movement disorder ataxia, which is characterized by impaired movement coordination affecting all body movements. In the arms, ataxia causes reaching movements with irregular, oscillating, and prolonged trajectory paths. People with cerebellar ataxia (PWCA) are also impaired in an important form of motor learning, called adaptation, which normally keeps movement well calibrated. In prior research, the principal investigator showed that PWCA can learn to correct their reaching movements if they instead employ reinforcement learning (RL). Although many PWCA learned optimally in RL conditions, this prior work found variability across individuals: some learned more than others. While adaptation critically relies on cerebellar integrity, RL depends more heavily on dopaminergic circuitry in the midbrain and excitatory plasticity in M1. Cerebellar damage has been shown to increase intracortical inhibition in M1, which may hamper the plasticity needed for RL. The repetitive TMS protocols of continuous theta burst stimulation (cTBS) and intermittent theta burst stimulation (iTBS) have further been shown to modulate intracortical inhibition: cTBS decreases it, while iTBS increases it. Here, the investigators will systematically test whether increased intracortical inhibition in M1 predicts RL capacity (Aim 1) and whether modulating inhibition in M1 can alter RL capacity in PWCA (Aim 2). 12 PWCA from a degenerative condition will complete 4 experimental sessions over a 6-month period. In session 1, TMS will be used to assess baseline recruitment curves for corticomotor excitability and short-interval intracortical inhibition, and the cortical silent period. PWCA will then complete a standardized clinical rating of their ataxia severity and an established behavioral task that requires learning a reaching skill using the RL paradigm. In sessions 2-4, PWCA will complete 3 additional sessions of the RL task. In each session, PWCA will receive cTBS, iTBS, or sham stimulation to modulate intracortical inhibition in M1 prior to performing the RL task. For Aim 1, the investigators will use multi-level regression to quantify relationships between TMS measures of M1 state and the magnitude and speed of learning in the RL task. For Aim 2, the investigators will use multi-level modeling to quantify differences in the magnitude and speed of learning across stimulation conditions. The investigators hypothesize that increased baseline inhibition in M1 will show a positive association with a lower magnitude and speed of learning in the RL task (Aim 1), and cTBS will improve the magnitude of learning, the speed of learning, or both, in the RL task relative to iTBS or sham stimulation (Aim 2).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebellar ataxia from cerebellar degeneration
* Normal or corrected-to-normal vision
* Normal or corrected-to-normal hearing
* Meet safety criteria for receipt of transcranial magnetic stimulation

Exclusion Criteria:

* Extrapyramidal signs on neurologic examination
* History of alcohol or illicit drug abuse
* Peripheral sensory loss in the arms
* Cognitive or attention deficits that interfere with testing, the capacity to understand and follow task instructions, or the capacity to provide informed consent
* Orthopedic injury or pain in the arms

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-12-19 (Estimated); Study Completion 2026-12-19 (Estimated)

PRIMARY OUTCOMES:
International Cooperative Ataxia Rating Scale Total Score | Baseline
  The sore out of 100 that results from assessment using the International Cooperative Ataxia Rating Scale (ICARS). The rating scale has a minimum score of 0 and a maximum score of 100. Higher scores indicate more severe impairment.
International Cooperative Ataxia Rating Scale Limb Coordination Sub-Score | Baseline
  The score out of 52 that results from assessment using the Limb Kinetic sub-section of the International Cooperative Ataxia Rating Scale (ICARS). The Limb Kinetic sub-score has a minimum score of 0 and a maximum score of 52. Higher scores indicate more severe impairment.
Reinforcement Learning Rate | During the intervention, assessed up to 10 days
  The slope of the time series of reach path lengths (determined from digital 3D kinematic data recorded using a motion capture system) over the first 80 trials of the intervention phase of the reinforcement motor learning task.
Total Reinforcement Learning | During the intervention, assessed up to 10 days
  The difference in mean reach path length (determined from digital 3D kinematic data recorded using a motion capture system) between the baseline phase and the end of the intervention phase of the reinforcement motor learning task.
Slope of the Corticomotor Excitability Recruitment Curve | Baseline
  The slope of motor evoked potential amplitudes (determined from electromyographic recordings of target muscle activity) between TMS intensities of 120-140% of resting motor threshold.
Slope of the Short-Interval Intracortical Inhibition (SICI) Recruitment Curve | Baseline
  SICI will be computed as the difference in average motor evoked potential amplitude (determined from electromyographic recordings of target muscle activity) between a TMS condition where a single conditioning pulse is applied 3 ms before a single test pulse and a TMS condition where only the test pulse is applied. A range of conditioning pulse TMS intensities will be tested and SICI will be measured for each. The outcome measure comprises the slope of the SICI values over each conditioning pulse intensity.
Cortical Silent Period | Baseline
  Single pulses of TMS will be applied at an intensity of 110% of resting motor threshold while participants tonically activate the target muscle at 20% of their maximum voluntary isometric contraction. 12 repetitions of the protocol will be performed. The outcome measure comprises the average time, in ms, from the end of the motor evoked potential to the reoccurrence of tonic background electromyographic activity.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda S Therrien, PhD, Principal Investigator — Moss Rehabilitation Research Institute
Locations (1):
- Moss Rehabilitation Research Institute, Elkins Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Participants will indicate, via written informed consent, whether they allow the study team to share the data collected as part of this study with other researchers. all individual participant data (IDP) that underlie results in a publication will be made available to other researchers. The study team will maintain the confidentiality of participant information to the extent possible. That is, participant's names and other identifying information will be removed from the data prior to sharing. The data will be coded with the participant's arbitrary study identification code. The key linking study identification codes to participant's identity will only be accessible to approved members of the study team.
Supporting Information: Analytic Code
Time Frame: Coded IPD data will be made available to other researchers immediately after publication, in compliance with the requirements of many academic journals in the motor control neuroscience field.
Access Criteria: Coded IPD and additional supporting information will be made available via a published repository on the Moss Rehabilitation Research Institute Sensorimotor Learning Laboratory Git Hub website. Requests for access to IPD will be reviewed by the study PI. Agreement to properly cite the original repository will be a requirement for approval of access.